CLINICAL TRIAL: NCT06668558
Title: Preemptive Treatment With Venetoclax Plus Azacitidine in Patients Diagnosed With Acute Myeloid Leukemia (AML) With Persistence or Reappearance of Measurable Residual Disease (MRD) After Frontline Chemotherapy and High-level MRD Prior to Allogeneic Hematopoietic Cell Transplantation (alloHCT)
Brief Title: Venetoclax + Azacitidine in Patients With Acute Myeloid Leukemia
Acronym: VERDI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CETLAM-LMA-AC-2024-01; 2024-510648-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: venetoclax; azacitidine; measurable residual disease (MRD); allogeneic hematopoietic cell transplantation (alloHCT)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: investigator-initiated, multicenter, multicohort, phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Patients diagnosed with a favorable ELN subtype AML, not intended for alloHCT in CR1, but who present an MRD failure by after frontline intensive chemotherapy, as defined in the 2021 update on MRD guidelines elaborated by the European LeukemiaNet MRD Working Party (Heuser et al. 2021)
  Interventions: Drug: Azacitidine (AZA); Drug: Venetoclax
- Cohort 2 (Experimental): Patients diagnosed with a non-favorable ELN AML subtype, intended to undergo alloHCT, in first complete morphological remission but harboring detectable MRD at time of alloHCT (>0.1%)
  Interventions: Drug: Azacitidine (AZA); Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine (AZA) — Dosing is 75 mg/m2 x 7 days (Q28days) After 2 courses, a first decision-making for allo-HCT based on bone marrow MRD assessment will be performed. After 4th course, a new MRD assessment will be performed.
  For cohort 1 treatment may continue up to cycle 12 (prioritized over allo-HCT). For cohort 2 treatment may continue up to cycle 24 (prioritizing allo-HCT)
Drug: Venetoclax — Dosing: 400 mg daily After 2 courses, a first decision-making for allo-HCT based on bone marrow MRD assessment will be performed. After 4th course, a new MRD assessment will be performed.
  For cohort 1 treatment may continue up to cycle 12 (prioritized over allo-HCT). For cohort 2 treatment may continue up to cycle 24 (prioritizing allo-HCT)

SUMMARY:
The VERDI study is an investigator-initiated, multicenter, multicohort, phase II trial with combination of venetoclax + azacitidine for patients treated for AML under according to an intensive chemotherapy protocol (CETLAM-20) failing to achieve or maintain MRD negativity at pre-established time-points: at chemotherapy completion for ELN favorable subtypes, and prior to alloHCT for non-favorable European LeukemiaNet (ELN) AML patients.

The primary objective is to determine Ven/Aza treatment activity in MRD clearance in patients diagnosed with AML with persistent MRD or MRD reappearance after frontline chemotherapy, or prior to alloHCT.

DETAILED DESCRIPTION:
The trial will enroll competitively between 25 and 29 patients.

Patients will be recruited in two independent cohorts depending on the pre-established time point for the intervention and ELN risk subtype:

Cohort 1: Patients diagnosed with a favorable ELN subtype AML, not intended for alloHCT in first complete remission (CR1), but who present an MRD failure by after frontline intensive chemotherapy, as defined in the 2021 update on MRD guidelines elaborated by the European LeukemiaNet MRD Working Party (Heuser et al. 2023):

In patients with persistent low-level MRD (<2%) after consolidation chemotherapy, an increase of MRD ≥1log10 between 2 positive samples Confirmed MRD conversion of MRD negativity to MRD positivity AML during subsequent follow-up (up to 3 years after chemotherapy completion

Cohort 2: Patients diagnosed with a non-favorable ELN AML subtype, intended to undergo alloHCT, in first complete morphological remission but harboring detectable MRD at time of alloHCT (>0.1%).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have confirmation of with acute myeloid leukemia (AML) with persistent measurable residual disease (MRD) or MRD reappearance after frontline intensive chemotherapy (including at least one cycle of cytarabine and anthracycline), and prior to allogeneic hematopoietic cell transplantation (allo-HCT).

   1. In patients with NPM1 mutation, qRT-PCR of NPM1 will be the method used to establish a molecular failure, defined as failure to achieve molecular response after consolidation therapy (NPM1mut/ABL1·100 > 0.1) or MRD reappearance after molecular response. All cases of molecular failure must be confirmed with a second MRD assessment in 2 to 4 weeks.
   2. In patients with core-binding factor AML, qRT-BCR of RUNX1-RUNX1T1 and CBFb-MYH11 transcripts will be used. Patients failing to achieve a major MRD reduction after consolidation therapy (i.e., RUNX1-RUNX1T1/ABL1·100>0.1 or CBFb-MYH11/ABL1·100>0.1), a log increase in MRD between two positive samples or confirmed MRD reappearance after molecular response will be considered as molecular failures and could be included in the trial.
   3. In the remaining cases, an appropriate leukemia-associated immunophenotype (LAIP) measured by multiparameter flow cytometry will be used for MRD surveillance. A cutoff of 0.1% will be used to define MRD positivity.
2. Age ≥18 years.
3. Without clinical signs of active central nervous system disease.
4. Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance status of ≤2 or Karnofsky performance status (KPS) equivalent.
5. Patients must have adequate renal function as demonstrated by a calculated creatinine clearance ≥ 30 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula.
6. Patients must have adequate liver function as demonstrated by:

   1. aspartate aminotransferase (AST) ≤ 3.0 × upper limit normal (ULN)
   2. alanine aminotransferase (ALT) ≤ 3.0 × ULN
   3. bilirubin ≤ 1.5 × ULN, unless due to Gilbert's syndrome
7. Non-sterile male patients must use contraceptive methods with partner(s) prior to beginning study drug administration and continuing up to 3 months after the last dose of study drug. Male patients must agree to refrain from sperm donation from initial study drug administration until 3 months after the last dose of study drug.
8. WOCBP must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting therapy; 2) throughout the entire duration of treatment; 3) during dose interruptions; and 4) for at least 6 months after discontinuation of therapy (last dose of study drug).
9. Patients must voluntarily sign and date an informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any research directed screening procedures.

Exclusion Criteria:

1. Patient has received other prior rescue treatment for MRD.
2. Patient is known to be positive for Human immunodeficiency virus (HIV) infection with the exception of those with an undetectable viral load under correct virological control throughout the study.

   Note: HIV testing is not required.
3. Patient is known to be positive for hepatitis B (HBV) or C (HCV) infection with the exception of those with an undetectable viral load.

   Note: Hepatitis B or C testing is not required and patients with serologic evidence of prior vaccination to HBV (i.e., HBsAg-, anti-HBs+ and anti-HBc-) may participate.
4. Patient has known active central nervous system (CNS) involvement from AML.
5. Patient has received within 7 days prior to the first dose of study drug: steroid therapy ≥ 20 mg/day (prednisone or equivalent) for antineoplastic intent; strong and moderate CYP3A inhibitors; strong and moderate CYP3A inducers.
6. Patient has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit within 3 days prior to the initiation of study treatment.
7. Patient has any history of clinically significant condition(s) that in the opinion of the investigator would adversely affect his/her participating in this study including, but not limited to:

   1. New York Heart Association heart failure > class 2.
   2. Renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or bleeding disorder independent of leukemia.
8. Patient has a malabsorption syndrome or other condition that precludes the enteral route of administration.
9. Patient exhibits evidence of uncontrolled systemic infection requiring therapy (viral, bacterial or fungal).
10. Patient has a history of other malignancies within the prior year to study entry, except for:

    1. Adequately treated in situ carcinoma of the breast or cervix uteri.
    2. Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin.
    3. Prostate cancer with no plans for therapy of any kind.
    4. Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
11. Pregnant and breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Rate of MRD conversion after 2 to 4 courses of study treatment | After the administration of 2 and 4 cycles (i.e. approximately 2 and 4 months after. Throughout the study period (up to 3 years) the initiation of study treatment)
  Defined as the percentage of patients who achieve MRD clearance after 2-4 courses of study treatment. Failure to achieve MRD negativity after 4 courses will be considered a treatment failure.

SECONDARY OUTCOMES:
Duration of MRD response | Throughout the study period, up to 3 years after chemotherapy completion. Throughout the study period (up to 3 years)
  Defined as the time elapsed from the first obtention of MRD clearance until MRD progression. Confirmed MRD conversion from MRD negativity to MRD positivity will be performed during subsequent follow-up.
Relapse risk after intervention | Throughout the study period, up to 3 years after chemotherapy completion. Throughout the study period (up to 3 years)
  Defined as the time elapsed from the intervention for AML until confirmed hematological relapse.
Safety profile | Throughout the study period, up to 3 years after chemotherapy completion. Throughout the study period (up to 3 years)
  Incidence of Treatment-Emergent Adverse Events Percentage of patients experiencing treatment-related adverse events (AEs).
Treatment Compliance | Throughout the study period, up to 3 years after chemotherapy completion. Throughout the study period (up to 3 years)
  Percentage of patients experiencing AEs that lead to dose modifications, including treatment interruption, delays and dose reductions.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Esteve, M.D.; Ph.D., Study Chair — Hematology department Institute Clínic of Hematological and Oncological diseases (ICMHO) Hospital Clínic of Barcelona
Locations (14):
- Spain (14):
  - University Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Institut Catala D oncologia Badalona, Badalona, Catalonia
  - Hospital Del Mar, Barcelona, Catalonia
  - Hospital De La Santa Creu I Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Vall D Hebron, Barcelona, Catalonia
  - Hospital Clinic De Barcelona, Barcelona, Catalonia
  - Institut Catala D oncologia Girona, Girona, Catalonia
  - Institut Catala D oncologia Hospitalet, L'Hospitalet de Llobregat, Catalonia
  - Hospital Universitari Arnau De Vilanova De La Gerencia Territorial De Lleida, Lleida, Catalonia
  - Hospital Universitari Joan XXIII De Tarragona, Tarragona, Catalonia
  - Fundacio Assistencial De Mutua De Terrassa, Terrassa, Catalonia
  - Hospital General Universitario Gregorio Maranon, Madrid, Madrid
  - Hospital Clinico Universitario De Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided
To protect confidentiality of patients the IPD will be restricted and only shared upon reasonable request if the purposes of this request complies with the conditions agreed with patients consent.